CLINICAL TRIAL: NCT05701423
Title: End of Dose Phenomena in Subcutaneous Natalizumab Treated MS Patients
Brief Title: A Study of End of Dose Phenomena in Subcutaneous Natalizumab Treated Multiple Sclerosis (MS) Participants
Acronym: SATURATE-MS
Status: Terminated | Type: Observational
Why Stopped: Due to low enrolment the sponsor decided to terminate the study
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: DE-TYS-12185
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Natalizumab (NTZ): Participants who receive NTZ intravenously (IV) or subcutaneously (SC) as standard interval dosing (SID), or as SC extended interval dosing (EID) will be followed prospectively for up to 30 weeks.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Administered as specified in the treatment arm.
  Other Names: Tysabri

SUMMARY:
The primary objective of this study is to better understand the pathophysiological background of end-of-dose symptoms (EOD) and thereby determine the percentage of participants who develop EOD under natalizumab (NTZ) as an example of interval therapy in MS and to detect specific changes through multimodal analyses, including radiological, blood and digital health measurements, that may be used as potential biomarkers in the future to map EOD.

DETAILED DESCRIPTION:
Participants will additionally be offered to record daily activity and sleep patterns as well as heart rate for the duration of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed Relapsing-Remitting Multiple Sclerosis (RRMS) according to 2017 revised McDonald criteria
* Initiation of treatment with SC NTZ according to summary of product characteristic (SmPC) and in accordance to national guidelines or
* Continuing treatment with IV NTZ
* Owns and be able to handle a smartphone

Key Exclusion Criteria:

* Participants with an acute MS relapse and/or a history of intravenous corticosteroid treatment within past six weeks
* Any comorbidity resulting in an impairment to understand or successfully complete the study such as (but not restricted to) psychiatric comorbidities or dementia
* Diagnosis of primary or secondary progressive MS
* Additional immunosuppression except of natalizumab

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include MS participants under NTZ therapy.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Develop End of Dose Symptoms (EOD) Under NTZ | Up to 30 weeks

SECONDARY OUTCOMES:
Change From Baseline in Expanded Disability Status Scale (EDSS) Score | Baseline up to 30 weeks
  The EDSS is used to quantify disability due to symptoms of MS and to track changes in disability status over time. Scores range from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). Higher scores indicate the worse level of disability.
Change From Baseline in Fatigue Scale for Motor and Cognitive Functions (FSMC) | Baseline up to 30 weeks
  Fatigue is rated using the self-administered 20-item FSMC questionnaire that includes ten questions related to motor fatigue and ten questions related to cognitive fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Minimum value is 20 (no fatigue at all) and maximum value is 100 (severe fatigue). Higher scores indicate higher fatigue.
Change From Baseline in Fatigue Severity Scale (FSS) | Baseline up to 30 weeks
  The FSS is a self-assessment questionnaire that provides a score as a measurement of the severity of fatigue. It consists of 9 questions scored from 1 to 7, low value indicates strong disagreement with the statement, whereas a high value indicates strong agreement. A total score of 36 or more suggests the presence of fatigue.
Change From Baseline in World Health Organization Quality of Life Brief Version (WHOQOL-BREF) Score | Baseline up to 30 weeks
  The WHOQOL-BREF questionnaire measures quality of life across 4 domains: Physical health, psychological health, social relationships and environment. It also includes one question on overall QOL and one on general health. The WHOQOL-BREF scores correlate highly (.89 or above) with WHOQOL-100 scores, and demonstrate good discriminant validity, content validity, internal consistency and test-retest reliability. The four WHOQOL-BREF domain scores will be used as main outcome measure. The measure is calculated by summing the point values for the questions corresponding to each domain and then transforming the scores to a 0-100 point interval, higher score correspond to greater QOL.
Change From Baseline in Brief Fatigue Inventory (BFI) Score | Baseline up to 30 weeks
  A questionnaire will be used to measure the severity of fatigue in the past 24 hours. This 9-item self-reported questionnaire is scored on a 0-10 numerical rating scale, where 0 and 10 represent absence and the highest severity of fatigue, respectively.
Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score | Baseline up to 30 weeks
  MSFC has 2 components: Timed 25-foot walk (T25FW) and 9-hole peg test (9HPT) [dominant and nondominant hands]. The MSFC Z-score is calculated by creating Z-scores for each component of the MSFC and averaging them to create an overall composite score. MSFC Z-score = (Z25-foot-walk + Z9HPT-2)/2, where Zj refers to Z-scores of component j. A Z-score represented the number of standard deviations participant's test result was higher (Z >0) or lower (Z <0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Klinik für Neurologie, Universitätsklinikum Düsseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/